CLINICAL TRIAL: NCT07401147
Title: Transcutaneous Electrical Stimulation for Pain Reduction During Labor: A Crossover Clinical Trial.
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Management During Labor: A Crossover Clinical Trial.
Acronym: TENS-LABOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Ricardo Arturo Gutierrez Ramirez, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PGO-UNAH-49-3-2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Labor Pain
Keywords: labor pain; Transcutaneous Electric Nerve Stimulation; Analgesia; Pain Management; Natural Childbirth
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, two-sequence (A-B, B-A), two-period crossover design. Sequence A: Active TENS first, then placebo. Sequence B: Placebo first, then active TENS. A 30-minute washout period between phases.
Who Masked: Participant, Outcomes Assessor
Masking Description: The TENS units for active and sham intervention are physically identical. A third party not involved in recruitment, intervention administration, or outcome assessment will pre-code all devices. Participants, the healthcare staff applying the devices, and the research staff assessing the primary outcome (pain via VAS) will be unaware of the device code (active/sham). The randomization list linking codes to sequences will be kept in a password-protected file accessible only to the study statistician until database lock. Blinding success will be formally assessed post-study via participant and staff questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS Intervention (Experimental): Participants receive transcutaneous electrical nerve stimulation (TENS) using the TENSCARE Perfect Mama+ unit. Electrodes are placed on the thoracolumbar region. The device is used for periods of 30-50 minutes every two hours during the active phase of labor (cervical dilation >=5 cm), or more frequently if desired by the participant.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); TENSCARE Perfect Mama+ TENS unit
- Sham/Placebo TENS (Sham Comparator): Participants undergo the same procedure with the TENS unit placed and electrodes attached, but the device remains switched off (no electrical stimulation is delivered)
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS); TENSCARE Perfect Mama+ TENS unit — A portable, dual-channel TENS unit (TENSCARE Perfect Mama+) delivering low to moderate intensity electrical currents via skin surface electrodes placed on the thoracolumbar region. It has three preset programs, 50-60 intensity levels, a BOOST button for contractions, and an open-circuit safety feature. Used for non-pharmacological labor pain relief.
  Arms: Active TENS Intervention
Device: Sham Comparator — Participants undergo the identical procedure with the TENS unit placed and electrodes attached in the same position, but the device remains switched off (no electrical stimulation is delivered).
  Arms: Sham/Placebo TENS

SUMMARY:
This is a randomized, double-blind, crossover clinical trial to evaluate the efficacy of transcutaneous electrical nerve stimulation (TENS) as a non-pharmacological therapeutic intervention for reducing pain in women during the active phase of labor. Nulliparous women with term pregnancies will be randomly assigned to sequences involving TENS intervention and placebo (device off) periods, separated by a washout. The primary outcome is labor pain intensity measured by the Visual Analog Scale (VAS). Secondary outcomes include duration of the active labor phase, maternal and neonatal safety profile, and childbirth experience satisfaction. The study will be conducted at the Hospital Escuela Universitario from feb 2026 to Ago 2026.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled, two-sequence, two-period crossover clinical trial. The study aims to evaluate the efficacy and safety of Transcutaneous Electrical Nerve Stimulation (TENS) as a non-pharmacological intervention for pain management during the active phase of first-stage labor.

The trial will be conducted in the Labor and Delivery Unit of the Maternal-Infant Block at Hospital Escuela Universitario in Tegucigalpa, Honduras. The unit is equipped with standard obstetric monitoring and care facilities.

Methodological Details:

Crossover Design: Each participant will act as her own control. Participants will be randomized to one of two sequences: 1) Active TENS followed by Sham TENS, or 2) Sham TENS followed by Active TENS.

Intervention & Control: The active intervention involves the use of a commercial, portable TENS unit (TENSCARE Perfect Mama+). The sham/placebo control involves the identical application of the device and electrodes but with the stimulator unit switched off. To maintain blinding, all devices will be visually identical and pre-coded by a third party not involved in data collection.

Washout Period: A standardized 30-minute washout period will be implemented between the active and sham phases. This duration is based on literature indicating the analgesic effects of TENS subside within 20-60 minutes post-use.

Intervention Periods: Each phase (active or sham) will have a defined application period during cervical dilation from ≥5 cm up to 10 cm. Pain assessments (Visual Analog Scale - VAS) will be conducted at baseline, 15 minutes, and 30 minutes after the initiation of each phase. The total duration of TENS/sham use per phase will be recorded.

Blinding Assessment: At the conclusion of the study, a blinding validation questionnaire will be administered to participants and clinical staff to assess the success of masking.

Additional Assessments: Beyond the crossover phases for pain measurement, the study will continue to observe participants in the experimental group to collect secondary data on the total duration of active labor, mode of delivery, maternal and neonatal complications, and postpartum satisfaction (using the Mackey Satisfaction Childbirth Rating Scale - MCSRS) within 24 hours after birth.

Statistical Considerations: The primary analysis will use linear mixed models or repeated measures ANOVA, accounting for treatment, period, and sequence effects. Carry-over effects will be specifically tested. The intention-to-treat (ITT) and per-protocol (PP) populations will be defined for analysis.

Scientific Rationale: The study design (crossover) increases statistical power and controls for inter-individual variability in pain perception. The double-blind, placebo-controlled approach minimizes bias. The protocol includes specific measures for bias minimization: centralized computerized randomization via REDCap, allocation concealment, and blinded outcome assessment.

Note: The full study protocol contains additional details on sample size calculation (n=132, based on a 1.0-point difference on VAS), safety monitoring, adverse event reporting, data management in REDCap, and ethical oversight by the Institutional Review Board of the Faculty of Medical Sciences, National Autonomous University of Honduras (UNAH).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.

Women aged 18-45 years.

Nulliparous.

Term singleton pregnancy (37-42 weeks).

Cephalic presentation.

Spontaneous onset of labor or induced/conducted labor under adequate control.

Cervical dilation of at least 5 cm at enrollment.

Normal amniotic fluid volume and reassuring fetal monitoring.

Uncomplicated pregnancy.

Exclusion Criteria:

* Multiple pregnancy.

Non-cephalic presentation.

Severe obstetric complications (e.g., preeclampsia, placental abruption).

Maternal chronic or acute diseases interfering with safety.

History of neurological/psychiatric disorders contraindicating TENS.

Abnormal fetal monitoring or amniotic fluid.

Pre-pregnancy BMI >30 kg/m².

Fetal demise.

Illiteracy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only pregnant womens are eligible
Enrollment: 132 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Labor Pain Intensity | Assessed at baseline (upon enrollment at >=5 cm dilation), at 15 minutes, and at 30 minutes after the start of each intervention phase (Active TENS or Sham) during the active phase of labor.
  Pain intensity during contractions, measured using the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Duration of Active Labor Phase | From study intervention start (>=5 cm) until delivery of the baby (up to 24 hours).
  Time elapsed from cervical dilation of 5 cm until complete cervical dilation (10 cm).
Maternal Satisfaction with Childbirth Experience | Assessed once within the first 24 hours postpartum (during the immediate puerperium, before hospital discharge).
  Satisfaction is measured using the validated Mackey Childbirth Satisfaction Rating Scale (MCSRS). This 35-item questionnaire uses a 5-point Likert scale (1 = Very Dissatisfied to 5 = Very Satisfied). The total score ranges from 35 to 175. A baseline score indicating satisfaction is considered to be ≥140 points (corresponding to an average rating of 4 or "Satisfied" across all items). Higher scores represent greater satisfaction with the childbirth experience. The scale assesses multiple dimensions including satisfaction with: the obstetrician, nursing staff, the newborn, the dilation phase, the expulsive phase, and overall comfort.

CONTACTS AND LOCATIONS:
Locations (2):
- Honduras (2):
  - Hospital Escuela, Tegucigalpa, Francisco Morazán Department
  - Instituto Hondureño de Seguridad Social, Tegucigalpa, Francisco Morazán Department

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data (IPD) available. The final decision will depend on the specific requirements of the target publication journal, further consultation with the local ethics committee regarding data sharing agreements, and a thorough assessment of our capacity to properly anonymize the data while preserving its scientific value for secondary analysis.

REFERENCES:
- [Background] Ge Z, He J, Zhang P, Zhao W, Zhu G, Zhang J, Song Z, Cui J, Jiang X, Yu W. Clinical Outcomes and Radiologic Parameters of Endoscopic Lumbar Interbody Fusion Using a Novel Nerve Baffle with a Minimum 1-year Follow-up. World Neurosurg. 2023 Aug;176:e181-e189. doi: 10.1016/j.wneu.2023.05.025. Epub 2023 May 12. PMID 37178917